CLINICAL TRIAL: NCT00589043
Title: Computed Tomography Laser Mammography Breast Imaging Device Model 1020
Brief Title: Computed Tomography Laser Mammography Breast Imaging Device
Acronym: CTLM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imaging Diagnostic Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: NA at present
Record Dates: First submitted 2007-12-24; First posted 2008-01-09 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the sensitivity and specificity of the CTLM system when used adjunctively with mammography compared to mammography alone in the heterogeneously and extremely dense breast population.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 21 and over
* Heterogeneously or extremely dense breast
* Schedule for biopsy
* Gave informed consent

Exclusion Criteria:

* Mammogram not performed within the last 60 days
* Open lesions on the breast
* Previous breast biopsy within 60 days of the CTLM scan
* Surgical deformity of breasts
* Commercial Tattoos
* Protoporphyria
* Lactating

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heterogeneous or extremely dense breast patient population scheduled for biopsy
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Jin, MD, Study Chair — Imaging Diagnostic Systems